CLINICAL TRIAL: NCT06157502
Title: Efficacy and Safety of Shuxuening Injection in the Treatment With Intravenous Thrombolysis in Patients With Ischemic Stroke: A Multicenter, Randomized, Double-blind, Placebo-parallel Controlled Trial
Brief Title: Shuxuening Injection in the Treatment With Intravenous Thrombolysis in Patients With Ischemic Stroke (SHINY)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Vice President, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HX-A-2023045
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Ischemic Stroke, Acute
Keywords: Ischemic Stroke; Intravenous Thrombolysis; Neuroprotective Therapy; Shuxuening Injection; Randomized Controlled Trial
MeSH Terms: conditions — Ischemic Stroke | interventions — shuxuening

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shuxuening injection (Experimental): Shuxuening Injection + Intravenous Thrombolysis
  Interventions: Drug: Shuxuening Injection
- Placebo (Placebo Comparator): Placebo + Intravenous Thrombolysis
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Shuxuening Injection — Receiving 20 ml Shuxuening injection plus 250ml 0.9% sodium chloride injection, intravenous drip once a day, for 10-14 days
  Arms: Shuxuening injection
Other: Placebo — Receiving 20 ml placebo Shuxuening injection plus 250ml 0.9% sodium chloride injection, intravenous drip once a day, for 10-14 days.
  Arms: Placebo

SUMMARY:
Shuxuening injection is a multi-target neuroprotective agent, it is expected to play a neuroprotective role on the basis of intravenous thrombolysis therapy. The primary purpose of this multicenter, randomized, double-blind, placebo-parallel controlled trial is to evaluate the efficacy and safety of Shuxuening injection in the treatment with intravenous thrombolysis in patients with ischemic stroke.

DETAILED DESCRIPTION:
Intravenous thrombolysis with rt-PA within the time window is the most effective drug for acute ischemic stroke, but there are still more than 50% patients with functional disability. Neuroprotective agents can reduce brain cell death after cerebral ischemia by blocking all links of ischemic cascade. Shuxuening injection is a multi-target neuroprotective agent, it is expected to play a neuroprotective role on the basis of intravenous thrombolysis therapy.

This study is a multicenter, randomized, double-blind, placebo-parallel controlled trial. A total of 1380 patients from 50 centers in China who could be treated within 6 hours of onset and have received or plan to undergo intravenous thrombolytic therapy will be enrolled and randomly assigned, in a 1:1 ratio, to receive Shuxuening injection (20 ml Shuxuening injection + 250 ml 0.9% sodium chloride injection), or to receive Shuxuening injection placebo (20 ml plus 250 ml 0.9% sodium chloride injection); both groups are treated for 10-14 days. The primary efficacy outcome is mRS Score 0 to 1 at 90 days, and the primary safety outcome is adverse events within 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older;
* Diagnosed with acute ischemic stroke;
* Within 6 hours of onset;
* Having received or plan to undergo intravenous thrombolytic therapy;
* NIHISS score of 4 to 25 points at enrollment;
* Signed informed consent.

Exclusion Criteria:

* mRS score greater than 1 point before the onset;
* Receiving neuroprotective agents, such as edaravone, edaravone dextrocamphorol, butylphthalein, etc. after the onset;
* Bleeding or other pathological brain disorders, such as vascular malformations, tumors, abscesses, or other common non-ischemic brain diseases (such as multiple sclerosis), detected by CT/MRI;
* History of clotting disorders, systemic bleeding, thrombocytopenia, or neutropenia;
* Severe hepatic or renal insufficiency (severe hepatic insufficiency refers to the ALT or AST levels above 3 times the upper limit of normal; severe renal insufficiency refers to the creatinine levels above 2 times the upper limit of normal);
* Allergic to Shuxuening injection or preparations containing ginkgo biloba (ginkgo biloba extract);
* Women who are pregnant or breastfeeding, and women of childbearing age who have a negative pregnancy test but refuse to take effective contraceptive measures;
* Participation in another clinical trial with an experimental product during the last 30 days;
* Other participants deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1380 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of mRS score 0 to 1 at 90 days after randomization | At 90 days after randomization
  The Modified Rankin Scale (mRS) score ranges from 0 to 6, with higher scores indicating worse functional outcome.

SECONDARY OUTCOMES:
The proportion of mRS score 0 to 2 at 90 days after randomization | At 90 days after randomization
  The Modified Rankin Scale (mRS) score ranges from 0 to 6, with higher scores indicating worse functional outcome.
The distribution of mRS scores at 90 days after randomization | At 90 days after randomization
  The Modified Rankin Scale (mRS) score ranges from 0 to 6, with higher scores indicating worse functional outcome.
NIHSS score improvement ≥4 points from baseline at 14 days after randomization or on discharge | At 14 days after randomization or on discharge
  The National Institutes of Health Stroke Scale (NIHSS) score ranges from 0 to 42, with higher scores indicating more severe neurological deficit.
EQ-5D score at 90 days after randomization | At 90 days after randomization
  The European Quality of Life 5-Dimension 3-Level (EQ-5D-3L) includes five dimensions. The sum score on each of the five dimensions ranges from 5 (all domains have level 1) to 15 (all domains have level 3), with higher scores indicating worse health-related quality of life.
The proportion of Barthel index score ≥95 points at 90 days after randomization | At 90 days after randomization
  The Barthel index score ranges from 0 to 100, with higher scores indicating greater independence.
Adverse events within 90 days after randomization | Within 90 days after randomization
Serious adverse events within 90 days after randomization | Within 90 days after randomization
Symptomatic intracranial hemorrhage (ECASS-III) within 90 days after randomization | Within 90 days after randomization
Symptomatic intracranial hemorrhage (SITS-MOST PH2) within 90 days after randomization | Within 90 days after randomization
All-cause death within 90 days after randomization | Within 90 days after randomization

CONTACTS AND LOCATIONS:
Locations (82):
- China (82):
  - Fangshan District First Hospital, Beijing, Beijing Municipality
  - Chongqing Nanchuan District People's Hospital, Chongqing, Chongqing Municipality
  - Chongqing Sanbo Chang'an Hospital, Chongqing, Chongqing Municipality
  - Chongqing Qianjiang Central Hospital, Qianjiang, Chongqing Municipality
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Heyuan People's Hospital, Heyuan, Guangdong
  - Huazhou People's Hospital, Maoming, Guangdong
  - Meizhou Hospital of Traditional Chinese Medicine, Meizhou, Guangdong
  - Yunfu People's Hospital, Yunfu, Guangdong
  - Wuchuan People's Hospital, Zhanjiang, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Wuming Hospital Affiliated to Guangxi Medical College, Nanning, Guangxi
  - Wuchuan Gelao and Miao Autonomous County Hospital of Traditional Chinese Medicine, Zunyi, Guizhou
  - Zunyi First People's Hospital, Zunyi, Guizhou
  - Baoding Xushui District People's Hospital, Baoding, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Wuchang Hospital of Traditional Chinese Medicine, Harbin, Heilongjiang
  - Puyang Anyang District Hospital, Anyang, Henan
  - Jiaozuo Coal Industry (Group) Co. Ltd. Central Hospital, Jiaozuo, Henan
  - Mengzhou Hospital of Traditional Chinese Medicine, Jiaozuo, Henan
  - Wenxian People's Hospital, Jiaozuo, Henan
  - Jiyuan Hospital of Traditional Chinese Medicine, Jiyuan, Henan
  - Kaifeng Central Hospital, Kaifeng, Henan
  - Lankao First Hospital, Kaifeng, Henan
  - Luohe Third People's Hospital, Luohe, Henan
  - Luoyang Yanshi People's Hospital, Luoyang, Henan
  - Pingdingshan First People's Hospital, Pingdingshan, Henan
  - Pingdingshan Second People's Hospital, Pingdingshan, Henan
  - Nanle Zhongxing Hospital, Puyang, Henan
  - Qinhuangdao Second Hospital, Qinhuangdao, Henan
  - Lingbao First People's Hospital, Sanmenxia, Henan
  - Shangqiu First People's Hospital, Shangqiu, Henan
  - Shangqiu Fourth People's Hospital, Shangqiu, Henan
  - Shangqiu Third Prople's Hospital, Shangqiu, Henan
  - Suixian Hospital of Traditional Chinese Medicine, Shangqiu, Henan
  - Suixian People's Hospital, Shangqiu, Henan
  - Xiayi People's Hospital, Shangqiu, Henan
  - Yongcheng Central Hospital, Shangqiu, Henan
  - Yongcheng People's Hospital, Shangqiu, Henan
  - Huixian People's Hospital, Xinxiang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Jingmen Hospital of Traditional Chinese Medicine, Jingmen, Hubei
  - Jingzhou First People's Hospital, Jingzhou, Hubei
  - Wuhan Central Hospital, Wuhan, Hubei
  - Wuhan Fifth Hospital, Wuhan, Hubei
  - Wuhan Hankou Hospital, Wuhan, Hubei
  - Wuhan Huangpi District People's Hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Liuyang Jili Hospital, Changsha, Hunan
  - Chenzhou First People's Hospital, Chenzhou, Hunan
  - Shaodong People's Hospital, Shaoyang, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technology, Baotou, Inner Mongolia
  - Tuquan People's Hospital, Hinggan, Inner Mongolia
  - Inner Mongolia Hangtian Hospital, Hohhot, Inner Mongolia
  - Zalantun Zhongmeng Hospital, Hulunbuir, Inner Mongolia
  - Zhalantun People's Hospital, Hulunbuir, Inner Mongolia
  - Huai'an Second People's Hospital, Huai'an, Jiangsu
  - Haicheng Hospital of Traditional Chinese Medicine, Anshan, Liaoning
  - Benxi Central Hospital, Benxi, Liaoning
  - Xinhua Hospital Affiliated to Dalian University, Dalian, Liaoning
  - Dandong Central Hospital, Dandong, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Shenyang First People's Hospital, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - Yan'an University Affiliated Hospital, Yan’an, Shaanxi
  - Ningjin People's Hospital, Dezhou, Shandong
  - Yuncheng People's Hospital, Heze, Shandong
  - Shandong Provincial Public Health Clinical Center, Jinan, Shandong
  - Guanxian People's Hospital, Liaocheng, Shandong
  - Linshu People's Hospital, Linyi, Shandong
  - Liaocheng Third People's Hospital, Liaocheng, Shangdong
  - Weihai Wendeng District People' Hospital, Weihai, Shangdong
  - Yantai Yeda Hospital, Yantai, Shangdong
  - Zibo Municipal Hospital, Zibo, Shangdong
  - Jincheng People's Hospital, Jincheng, Shanxi
  - Yuci District People's Hospital, Jinzhong, Shanxi
  - Linfen Central Hospital, Linfen, Shanxi
  - Linfen People's Hospital, Linfen, Shanxi
  - Tianjin Xiqing Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Shihezi University Medical College, Shihezi, Xinjiang
  - Yunnan Third People's Hospital, Kunming, Yunnan